CLINICAL TRIAL: NCT05283382
Title: Cannabidiol Effects on Learning and Anxiety
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Robert Astur, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: H21-0159
Record Dates: First submitted 2022-02-23; First posted 2022-03-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Anxiety and Fear
Keywords: social anxiety; fear conditioning; cannabidiol; electrodermal response
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Drug group vs. Placebo group
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): 600 mg Cannabidiol Isolate Gel Capsules / participant. One-time dose.
  Interventions: Drug: Cannabidiol Oral Product
- Placebo (Placebo Comparator): Same number of placebo capsules / participant. One-time dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabidiol Oral Product — Participants will receive a one-time dose of 600 mg Cannabidiol Isolate Gel Capsules in the form of six 100mg capsules.
  Arms: Cannabidiol
Other: Placebo — Participants will receive a one-time dose of placebo capsules in the form of six capsules.
  Arms: Placebo

SUMMARY:
To examine the extent to which Cannabidiol (CBD) enhances fear conditioning extinction in college undergraduates who show elevated social anxiety. Undergraduates who display elevated social anxiety on standard assessments will be recruited at the University of Connecticut. All participants will be put in a standard fear conditioning paradigm where they are conditioned to fear a face that occasionally is followed by a shock to their wrist. The other face never is paired with a shock. After everybody learns this, half of the participants will receive 600 mg CBD Isolate Gel Capsules one time, and the other half will receive a placebo dose. Participants will then be presented with the faces with no shocks, and the rate and duration of extinction as measured by electrodermal response as well as subjective fear ratings via a visual analogue scale will be examined. It is hypothesized that participants that receive CBD will display enhanced extinction compared to the placebo group, as evidenced by reduced electrodermal response and reduced visual analogue fear ratings.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age

Exclusion Criteria:

1. Difficulties seeing a computer screen
2. Anyone currently taking CBD within the last 24 hours.
3. Anyone using any cannabis product within the last 24 hours.
4. Heart problems or heart disease
5. A neurological disorder such as epilepsy, stroke, multiple sclerosis, tumor, vascular malformations, aneurysm
6. Are currently pregnant or breast-feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Electrodermal activity | 20 minutes
  Electrodermal response as measured by galvanic skin response electrodes that are attached to two of the fingers via sticker electrodes. These passively measure the conductance of the sweat glands on the fingers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No